CLINICAL TRIAL: NCT06357260
Title: Evaluation of Efficacy of Pregabalin as an Add on Therapy With Carbamazepine in Patients of Trigeminal Neuralgia"- A Randomized Control Trial
Brief Title: Pregabalin as an add-on Therapy to Carbamazepine in Trigeminal Neuralgia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shifa OMR
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Pregabalin; Carbamazepine; Control Groups

STUDY DESIGN:
Intervention Model Description: Test group-1 will be administered carbamazepine+pregabalin with fixed dose of pregabalin 75mg BD and carbamazepine being titrated as per patients's need and follow up done after 1 week with subsequent follow up at 2,4,6 and 8 weeks.
  control group all the armamentarium and procedure will remain same except that dose titration of carbamazepine is done till patient is relieved of pain.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group-1 (Experimental): Carbamazepine+pregabalin with fixed dose of pregabalin 75mg BD and carbamazepine being titrated as per patients's need
  Interventions: Drug: Pregabalin and Carbamazepine
- Control group (Active Comparator): Carbamazepine with dose of Carbamazepine being titrated as per patients's need
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Pregabalin and Carbamazepine — Carbamazepine+pregabalin with fixed dose of pregabalin 75mg BD and carbamazepine being titrated as per patients's need
  Other Names: Test group
  Arms: Test group-1
Drug: Carbamazepine — Carbamazepine with dose of Carbazmaepine being titrated as per patients's need
  Other Names: Control group
  Arms: Control group

SUMMARY:
Trigeminal neuralgia is a very painful condition associated with paroxysmal severe episodes of pain. Carbamazepine has been the first line of drug for Trigeminal Neuralgia. However, there are several adverse effects linked with Carbamazepine like drowsiness, accommodation disorders, hepatitis, derangement in hepatic enzymes, renal dysfunction. Pregabalin which is an established drug in neuropathic pain has better pharmacokinetic nature which allows for easy management and rapid dose escalation to therapeutic doses. There have been only few trials evaluating efficacy of Pregabalin in classical trigeminal neuralgia. Thus, the present study is designed to evaluate the efficacy of Pregabalin as an add-on therapy to carbamazepine in patients suffering from Trigeminal Neuralgia. In present trial 50 patients fulfilling the exclusion and inclusion criteria will be recruited in two arms that is test group and the control group. The test group will be prescribed carbamazepine along with fixed dose of Pregabalin 75mg twice daily while the control group will be prescribed carbamazepine only. The dose of carbamazepine will be titrated in both groups as per patients need. The outcome regarding pain relief, quality of life and adverse effects and mean dose of carbamazepine required in both groups will be evaluated.

DETAILED DESCRIPTION:
AIM

Evaluation of Efficacy of Pregabalin as an add on therapy with Carbamazepine in patients with trigeminal neuralgia.

OBJECTIVES

Primary objectives-

1. To compare the change in pain intensity in both groups.

Secondary objectives-

1. To evaluate the mean dose of carbamazepine used in both the groups.
2. To evaluate quality of life.
3. To evaluate the patient satisfaction in both groups.
4. To evaluate the need for additional pain medicine in both groups.

STUDY DESIGN

A randomized clinical trial will be conducted in department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.

STUDY SETTING

Hospital based study - Patients diagnosed with Trigeminal neuralgia will be recruited in study from regular OPD of the department of Oral Medicine and Radiology.

STUDY PERIOD

This study will be completed in 1 year.

STUDY SUBJECTS

Patients diagnosed with classical Trigeminal neuralgia will be recruited in the study from regular OPD of the Department of Oral Medicine and Radiology, PGIDS, Rohtak, Haryana. A total of 50 patients would compromise; Test group (n=25) and Control group (n=25).

METHOD OF RECRUITMENT Patient will be randomly allocated to test and control groups by using simple random sampling.

INTERVENTION

Clinically and MRI proven cases of classical Trigeminal neuralgia will be randomly and equally divided into test group and control group. The selected subjects will be divided into two groups.

TEST GROUP

Test group will be administered carbamazepine+pregabalin with fixed dose of pregabalin 75mg BD and carbamazepine being titrated as per patients's need and follow up done after 1 week with subsequent follow up at 2,4,6 and 8 weeks.

CONTROL GROUP

In control group all the armamentarium and procedure will remain same except that dose titration of carbamazepine is done till patient is relieved of pain.

Both groups will be assessed for the following parameters: intensity of pain, at the baseline ,1st week, 2nd week, 4th week ,6th week and 8th weeks interval.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients diagnosed with Trigeminal neuralgia with classical types without concomitant pain as per ICHD-II.
* Patient's consent for participation in this study.

EXCLUSION CRITERIA

* Pregnant and lactating women
* Patients on anti-depressants like sodium valproate
* History of excessive alcohol intake
* Hepatic or renal insufficiency
* Known tolerance/allergy to study drug
* Non -compliant during screening period
* Any other hepatic microsomal enzyme inhibitors (to avoid risk for toxicity)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 0-8 weeks
  0- no pain 10-worst pain possible .Higher score means worst outcome
Brief pain inventory | 0-8 weeks
  1-4=mild pain. 07-10 =severe pain. Higher score means worst outcome

SECONDARY OUTCOMES:
Mean dose of carbamazepine | 0-8 weeks
  lower dose requirement of carbamazepine means better outcome
Patient global impression of scale | 0-8 weeks
  1- very much improved and 7-very much worse .Higher score means worst outcome
Liverpool scale | 0-8 weeks
  Scale meant for adverse events score ranging from 19 -76 with higher score indicating greater adverse event related to drug

CONTACTS AND LOCATIONS:
Overall Officials: Shifa Akhtar, BDS, Principal Investigator — Post Graduate Institute of Dental Sciences ,Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No